CLINICAL TRIAL: NCT00739102
Title: S.M.A.R.T.® Nitinol Self-Expandable Stent in the Treatment of Obstructive Superficial Femoral Artery Disease (STROLL)
Brief Title: S.M.A.R.T.® Nitinol Self-Expandable Stent in the Treatment of Obstructive Superficial Femoral Artery Disease
Acronym: STROLL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05-6201
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Results first posted 2013-09-18 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Superficial Femoral Artery Disease
Keywords: Superficial Femoral Artery; Nitinol Self-Expandable Stent System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): S.M.A.R.T.® Nitinol Self-Expandable Stent System
  Interventions: Device: S.M.A.R.T. ® Stent

INTERVENTIONS:
Device: S.M.A.R.T. ® Stent — The Cordis S.M.A.R.T.® Nitinol Stent System is a self-expandable, crush recoverable stent with a diameter larger than that of the arterial lumen. The stent is indicated for use in a vessel with a diameter 1 to 2 mm smaller than the nominal stent diameter. This stent will open to the diameter of the artery and will continue to apply expanding force on the artery.

SUMMARY:
A multi-center, non-randomized, single-arm, prospective trial evaluating the safety and effectiveness of the S.M.A.R.T.™ Nitinol Stent System implantation in approximately 250 patients with obstructive superficial femoral artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 30 years
* For women of child bearing potential, a pregnancy test within 7 days prior to index procedure (the test results must be negative to be eligible).
* Symptomatic leg ischemia by Rutherford/Becker Classification (category 2, 3 or 4) with a resting or exercise ABI </= 0.8.
* A single superficial femoral artery lesion with > 50% stenosis or total occlusion.
* Stenotic lesion or occluded length within the same vessel (one long or multiple serial lesions) >/= 4.0 cm to </= 15.0 cm, by visual estimate. The stenosis must be treatable with no more than two stents, minimizing the stent overlap whose combined length </= 170 mm.
* Reference vessel diameter (RVD) >/= 4.0 mm and </= 6.0 mm by visual assessment.
* All lesions are to be located at least three centimeters proximal to the superior edge of the patella.
* Patent infrapopliteal and popliteal artery, i.e., single vessel runoff or better with at least one of three vessels patent (< 50% stenosis) to the ankle or foot.
* The guidewire is across the target lesion(s) and located intraluminally within the distal vessel.
* Poor aortoiliac or common femoral "inflow" (i.e. angiographically defined > 50% stenosis of the iliac or common femoral artery) that would be deemed inadequate to support a femoropopliteal bypass graft must be successfully treated prior to treatment of the target lesion. This can be done just prior to treatment of the target lesion. Successful treatment is defined as <30% stenosis after either PTA or stenting of the inflow lesion. After treatment of the inflow lesion, if the peak to peak pressure gradient across the inflow lesion is </= 20mmHg and the peak to peak pressure gradient across the SFA target lesion is >/= 20mmHg, then the patient will be included in the study.
* A patient with bilateral obstructive SFA disease is eligible for enrollment into the study.
* Eligibility for standard surgical repair, if necessary.
* A patient who requires a coronary intervention, should have it performed at least 7 days prior to the treatment of the target lesion.
* Patient or authorized representative must provide written informed consent and written HIPAA authorization prior to initiation of study procedures.
* Patient must be willing to comply with the specified follow-up evaluation schedule.

Exclusion Criteria:

* Thrombophlebitis, uremia, or deep venous thrombus, within past 30 days.
* Receiving dialysis or immunosuppressant therapy.
* Thrombolysis of the target vessel within 72 hours prior to the index procedure where complete resolution of the thrombus was not achieved.
* Recent stroke within past 90 days.
* Femoral, iliac or aortic aneurysm or aneurysm in the SFA or popliteal artery within past 5 years.
* Required stent placement via a popliteal approach.
* Required stent placement across or within 0.5 cm of the SFA / PFA bifurcation.
* Procedures which are pre-determined to require stent-in-stent placement to obtain patency, such as severe calcification which is resistant to stenting, or for in-stent restenosis.
* Significant vessel tortuosity or other parameters prohibiting access to the lesion or 90° tortuosity which would prevent delivery of the stent device.
* Previously deployed stent within the SFA of the target limb.
* Known allergies to the following: aspirin, clopidogrel bisulfate (Plavix®) or ticlopidine (Ticlid®), heparin, Nitinol (nickel titanium), contrast agent, that cannot be medically managed.
* Presence of thrombus prior to crossing the lesion
* Tissue loss due to ischemic disease (Rutherford/Becker category 5 or 6)
* Serum creatinine level >/= 2.5 mg/dl at time of screening visit
* Known or suspected active infection at the time of the procedure
* Bleeding diathesis
* Presence of an aortic, iliac or femoral artificial graft
* Life expectancy less than one year, or any other factors preventing clinical followup.
* Use of cryoplasty, laser, or atherectomy devices on the target vessel at the time of index procedure
* In-stent restenotic lesions at time of procedures.
* Restenotic lesion that had previously been treated by atherectomy, laser, or cryoplasty within 90 days of the index procedure.
* Patient is unwilling or unable to comply with procedures specified in the protocol or has difficulty or inability to return for follow-up visits as specified by the protocol.
* Patient is known to be pregnant, incarcerated, mentally incompetent, and/or alcohol or drug abuser.
* Patient is currently participating in any other investigational drug or medical device study that has not completed primary endpoint(s) evaluation or clinically interferes with the endpoints from this study or future participation in such studies prior to the completion of this study.
* Patient has had major surgical or interventional procedures unrelated to this study within 30 days prior to this study or planned surgical or interventional procedures within 30 days of entry into this study. Interventional procedures performed to the ipsilateral iliac artery to provide access will be allowed.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-08; Primary Completion 2011-05 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Gray, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 250 patients were enrolled from August 14, 2008 to March 15, 2010 across 39 clinical sites in the U.S.
Pre-assignment Details: This is a multi-center, non-randomized, single-arm, prospective trial. Patients were eligible for enrollment if they met all inclusion criteria and none of the exclusion criteria.
Groups:
- S.M.A.R.T.® Nitinol Stent System: The Cordis S.M.A.R.T. ®Nitinol Stent System is a self-expandable, crush recoverable stent with a diameter larger than that of the arterial lumen. The stent is indicated for use in a vessel with a diameter 1 to 2 mm smaller than the nominal stent diameter. This stent will open to the diameter of the artery and will continue to apply expanding force on the artery.
Period: Overall Study
Arm/Group | S.M.A.R.T.® Nitinol Stent System
Started | 250
Completed | 235 (Completed 12-Month Follow-up)
Not Completed | 15
Not completed — Death | 5
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Population: Modified Intent-To-Treat (ITT) Population
Groups:
- S.M.A.R.T.™ Nitinol Stent System: The Cordis S.M.A.R.T.™ Nitinol Stent System is a self-expandable, crush recoverable stent with a diameter larger than that of the arterial lumen. The stent is indicated for use in a vessel with a diameter 1 to 2 mm smaller than the nominal stent diameter. This stent will open to the diameter of the artery and will continue to apply expanding force on the artery.
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 93
  >=65 years | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.71 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 240
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 0
  Asian | 1
  Black or African American | 31
  Native Hawaiian or Other Pacific Islander | 0
  White or Caucasian | 214
  Middle Eastern | 1
  Hispanic | 3
  Other | 0
Region of Enrollment [Number; unit: participants]
  United States | 250

OUTCOME MEASURES:

1. Primary Outcome: 12-month Primary Patency Rate
Description: Primary patency is defined as no significant reduction of flow detectable by Duplex ultrasound through the index lesion and no further clinically driven target vessel revascularization performed in the interim. Significant reduction of flow is binary restenosis defined as the diameter stenosis >50% with a peak systolic velocity ratio >2.0 as measured by Duplex ultrasound.
Time Frame: 12 months
Population: As a subset of the modified ITT, this analysis population consisted of the subjects who had ultrasound assessment at 12 months or had target vessel revascularization (TVR) performed by 12 months.
Measure: Number; unit: participants
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 215
participants
  Subjects Achieved Primary Patency | 143 [lower limit 60]
  Subjects Didn't Achieve Primary Patency | 72
Statistical Analysis 1: Comparison: S.M.A.R.T.™ Nitinol Stent System; The null hypothesis to be tested was Ho: P = 0.66 against Ha: P > 0.66, where 0.66 was the Objective Performance Criteria (OPC). A sample size of 212 subjects was required to achieve 90% power to reject the 66% 12-months patency rate at a one-sided 2.5% significance level when the unknown true patency is at 76%; Test type: Superiority or Other; p = 0.437, Agresti-Coull method — The observed rate of primary patency at 12 month was 66.5% (143/215) with a lower 95% confidence interval of 60.0%; Proportion - 12-month patency rate = 0.665, 95% CI 2-sided [0.6 to 0.725], Standard Error of Mean 0.032 — The 95% confidence intervals and the standard error were calculated using the Agresti-Coull method

2. Secondary Outcome: Death Rate at 30-day Post Procedure
Time Frame: 30 days
Population: Active subjects in the Modified ITT population at 30-day post procedure
Measure: Number; unit: participants
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 248
participants | 0

3. Secondary Outcome: Death at 12-month Post Procedure
Time Frame: 12 months
Population: Active subjects in the Modified ITT population at 12-month post procedure
Measure: Number; unit: participants
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 236
participants | 5
Statistical Analysis 1: Comparison: S.M.A.R.T.™ Nitinol Stent System; Test type: Superiority or Other; Death Rate (%) = 2.1, 95% CI 2-sided [0.7 to 4.9]

4. Secondary Outcome: Index Limb Amputation at 30-day Follow up
Description: Index Limb Amputation is defined as surgical removal of all or part of the lower extremity from the toe up.
Time Frame: 30 day
Population: Active subjects in the Modified ITT population at 30 days post procedure
Measure: Number; unit: participants
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 248
participants | 0
Statistical Analysis 1: Comparison: S.M.A.R.T.™ Nitinol Stent System; Test type: Superiority or Other; Index Limb Amputation Rate (%) = 0.0, 95% CI 2-sided [0.0 to 1.5]

5. Secondary Outcome: Clinically Driven Target Vessel Revascularization (TVR) at 30-day Post Procedure
Description: A clinically driven TVR is any intervention of the target vessel following documented recurrent symptomatic leg ischemia by Rutherford/Becker Classification (category 2, 3 or 4), with a resting or exercise Ankle-Brachial Index (ABI) ≤ 0.8 and >50% diameter in-lesion stenosis by angiography. Revascularization of a target vessel with an in-lesion diameter stenosis of >70% by angiography, in the absence of the previously mentioned ischemic signs or symptoms, will also be considered clinically driven.
Time Frame: 30 days
Population: Active subjects in the Modified ITT population at 30-day post procedure
Measure: Number; unit: participants
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 248
participants | 0
Statistical Analysis 1: Comparison: S.M.A.R.T.™ Nitinol Stent System; Test type: Superiority or Other; Clinically Driven TVR Rate (%) = 0.0, 95% CI 2-sided [0.0 to 1.5]

6. Secondary Outcome: Clinically Driven Target Vessel Revascularization (TVR) at 12-month Post Procedure
Description: as for outcome 5
Time Frame: 12 months
Population: Active subjects in the Modified ITT population at 12-month post procedure
Measure: Number; unit: participants
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 236
participants | 32
Statistical Analysis 1: Comparison: S.M.A.R.T.™ Nitinol Stent System; Test type: Superiority or Other; Clinically Driven TVR Rate (%) = 13.6, 95% CI 2-sided [9.5 to 18.6]

7. Secondary Outcome: Stent Fracture at 12-month Follow Up
Description: Stent fracture was assessed by x-ray evaluation.
Time Frame: 12 months
Population: Active subjects in the Modified ITT population at 12-month post procedure
Measure: Number; unit: participants
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 197
participants | 3
Statistical Analysis 1: Comparison: S.M.A.R.T.™ Nitinol Stent System; Test type: Superiority or Other; Stent Fracture Rate (%) = 1.5, 95% CI 2-sided [0.3 to 4.4]

8. Secondary Outcome: Index Limb Ischemia at 6-month Follow up
Description: Index Limb Ischemia is defined by Rutherford/Becker Classification categories 3 through 6.
Time Frame: 6 months
Population: Active subjects in the Modified ITT population at 6-month post procedure
Measure: Number; unit: participants
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 215
participants | 12
Statistical Analysis 1: Comparison: S.M.A.R.T.™ Nitinol Stent System; Test type: Superiority or Other; Index Limb Ischemia Rate (%) = 5.6

9. Primary Outcome: Primary Safety Endpoint
Description: Primary safety endpoint is defined as the rate of freedom from all causes of death, index limb amputation, and clinically driven target lesion revascularization (TLR) through 30 days. A clinically driven TLR is any intervention in the stented target lesion following documented recurrent symptomatic leg ischemia by Rutherford/Becker Classification (category 2, 3 or 4), with a resting or exercise ABI ≤ 0.8 and >50% diameter in-lesion stenosis by angiography. Revascularization of a target lesion with an in-lesion diameter stenosis of >70% by angiography, in the absence of the previously mentioned ischemic signs or symptoms, will also be considered clinically driven.
Time Frame: 30 days
Population: Active subjects in the Modified ITT population at 30 days post procedure
Measure: Number; unit: participants
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 248
participants
  Subjects Achieved Primary Safety Endpoint | 248
  Subjects Didn't Achieve Primary Safety Endpoint | 0
Statistical Analysis 1: Comparison: S.M.A.R.T.™ Nitinol Stent System; The null hypothesis to be tested was Ho: P = 0.88 against Ha: P > 0.88, where 0.88 was the Objective Performance Criteria (OPC); Test type: Superiority or Other; p < 0.001, Agresti-Coull method; Primary safety endpoint rate (%) = 100, 95% CI 2-sided [98.2 to 100]

10. Secondary Outcome: Index Limb Ischemia at 12-month Follow up
Description: Index Limb Ischemia is defined by Rutherford/Becker Classification categories 3 through 6.
Time Frame: 12 months
Population: Active subjects in the Modified ITT population at 12-month post procedure
Measure: Number; unit: participants
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 214
participants | 18
Statistical Analysis 1: Comparison: S.M.A.R.T.™ Nitinol Stent System; Test type: Superiority or Other; Index Limb Ischemia Rate (%) = 8.4

11. Secondary Outcome: Rutherford/Becker Classification at 30-day Follow Up
Description: The Rutherford/Becker Classification is a commonly used clinical staging system which allows clinicians to describe and discuss patients with peripheral artery disease. The classification has seven stages as follows:
  1. Stage 0 - Asymptomatic, no hemodynamically significant occlusive disease
  2. Stage 1 - Mild claudication
  3. Stage 2 - Moderate claudication
  4. Stage 3 - Severe claudication
  5. Stage 4 - Ischemic rest pain
  6. Stage 5 - Minor tissue loss, non-healing ulcer, focal gangrene with diffuse pedal ischemia
  7. Stage 6 - Major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable
Time Frame: 30 days
Population: Active subjects in the Modified ITT population at 30-day post procedure
Measure: Number; unit: participants
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 243
participants
  Rutherford/Becker Classification - 0 | 157
  Rutherford/Becker Classification - 1 | 39
  Rutherford/Becker Classification - 2 | 38
  Rutherford/Becker Classification - 3 | 8
  Rutherford/Becker Classification - 4 | 1
  Rutherford/Becker Classification - 5 | 0
  Rutherford/Becker Classification - 6 | 0

12. Secondary Outcome: Rutherford / Becker Classification Category at 12-month Follow Up
Time Frame: 12 months
Population: Active subjects in the Modified ITT population at 12-month post procedure
Measure: Number; unit: participants
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 214
participants
  Rutherford/Becker Classification - 0 | 125
  Rutherford/Becker Classification - 1 | 39
  Rutherford/Becker Classification - 2 | 32
  Rutherford/Becker Classification - 3 | 16
  Rutherford/Becker Classification - 4 | 1
  Rutherford/Becker Classification - 5 | 1
  Rutherford/Becker Classification - 6 | 0

13. Secondary Outcome: Major Adverse Events at 12-month Post Procedure
Description: Major adverse events included death, index limb ischemia, index limb amputation, clinically driven TLR, and significant embolic events, which were defined as causing end-organ damage.
Time Frame: 12 months
Population: Active subjects in the Modified ITT population at 12-month post procedure
Measure: Number; unit: participants
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Number analyzed (Participants) | 236
participants | 34
Statistical Analysis 1: Comparison: S.M.A.R.T.™ Nitinol Stent System; Test type: Superiority or Other; Major adverse event rate (%) = 14.4, 95% CI 2-sided [10.2 to 19.5]

ADVERSE EVENTS:
Arm/Group | S.M.A.R.T.™ Nitinol Stent System
Serious Adverse Events (participants affected / at risk) | 5/250
Other Adverse Events (participants affected / at risk) | 93/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S.M.A.R.T.™ Nitinol Stent System (N=250)
Death (General disorders) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S.M.A.R.T.™ Nitinol Stent System (N=250)
Arterial restenosis (Injury, poisoning and procedural complications) | 3 (3)
Catheter site haematoma (Injury, poisoning and procedural complications) | 5 (5)
Catheter site haemorrhage (Injury, poisoning and procedural complications) | 4 (4)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 48 (56)
Stent occlusion (Injury, poisoning and procedural complications) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10)
Femoral artery dissection (Vascular disorders) | 5 (5)
Intermittent claudication (Vascular disorders) | 17 (20)
Peripheral ischaemia (Vascular disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days